CLINICAL TRIAL: NCT01460238
Title: Lipoprotein Lipase Expression in Chronic Lymphocytic Leukemia
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Frederick Lansigan, Assistant Professor of Medicine, Dartmouth-Hitchcock Medical Center
Other Study IDs: D11065
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Lipoprotein Lipase; Chronic Lymphocytic Leukemia; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10 cc of peripheral blood and Archived lymph node tissue or bone marrow samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No treatment: No intervention. Each patient will have blood drawn at a standard of care venipuncture.

SUMMARY:
The investigators hypothesize that Lipoprotein Lipase (LPL) expression on Chronic Lymphocytic Leukemia (CLL) cells will predict a more aggressive clinical course. The results from this proposal will validate the use of a novel antibody developed at Dartmouth-Hitchcock in CLL and will predict CLL patients that have a more aggressive form of the disease. The investigators work will also provide direct evidence that LPL is expressed on CLL cells and provides a critical source of fatty acids required by the CLL cells to grow and survive. Fatty acid metabolism may become a therapeutic target in CLL in the future.

DETAILED DESCRIPTION:
The investigators plan to use a novel antibody developed at Dartmouth-Hitchcock Medical Center to characterize the expression of LPL in CLL. Peripheral blood from CLL patients will be analyzed by flow cytometry to detect the expression of LPL and to investigate if LPL expression correlates with a more aggressive type of CLL. The investigators propose that LPL protein expression on CLL cells is prognostic and that LPL and other proteins involved in fatty acid metabolism are critical for CLL cells to survive.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL as per National Cancer Institute Working Group Guidelines
* Patients undergoing routine blood draws as part of their ongoing follow up for CLL
* 18 years or older
* Ability to provide consent in English
* Patient must have measurable disease as defined by an absolute lymphocyte count greater than 5,000/mm3 or have archived lymph node or bone marrow with CLL involvement.

Exclusion Criteria:

* Patients who have received cytotoxic drug, oral or intravenous steroid or targeted antibody therapy for their CLL,
* other hematologic malignancy or other disease process within the past 6 months are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Dartmouth-Hitchcock Medical Center's Norris Cotton Cancer Center with CLL
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2011-10; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
LPL Protein Expression | 1 year
  Determine the degree of LPL protein expression in CLL cells using a novel LPL antibody, correlate with IgHV mutation status, and compare this association with other prognostic markers

SECONDARY OUTCOMES:
Fatty acid acquisition and synthesis | 1 year
  Demonstrate that CLL cells also possess the enzymatic machinery for fatty acid acquisition and synthesis as shown by the expression of LPL, CD36, SDC1, and fatty acid synthase

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Lansigan, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States